CLINICAL TRIAL: NCT03939052
Title: Protein Requirements in Phenylketonuria (PKU) Patients Compared Using PKU Sphere™ | Glycomacropeptide (GMP) and an L-amino Acid-based Product
Brief Title: Protein Requirements in Adults With Phenylketonuria (PKU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vitaflo International, Ltd (Industry)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H18-03464
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Phenylalanine metabolism; Protein requirements; Indicator Amino acid Oxidation; Stable isotopes; GMP; Glycomacropeptide
MeSH Terms: conditions — Phenylketonurias | interventions — caseinomacropeptide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein intake (Experimental): Free amino acids vs. Glycomacropeptide (GMP)
  Interventions: Dietary Supplement: Free amino acids intake

INTERVENTIONS:
Dietary Supplement: Free amino acids intake — Oral consumption of eight hourly experimental meals- -4 tracer free experimental meals containing a mixture of free amino acids and calories from protein free flavoured liquid, protein free cookies and corn oil -4 isotopically labeled experimental meals. The same protocol will be repeated with glycomacropeptide (GMP).
  Other Names: glycomacropeptide (GMP) intake

SUMMARY:
Phenylketonuria (PKU) is an inherited inborn error of phenylalanine (PHE) metabolism caused by decreased activity of phenylalanine hydroxylase (PAH) enzyme. Therefore, PHE accumulates in plasma leading to mental problems. Treatment is a phenylalanine-restricted diet with sufficient protein. However, the optimum protein requirements are still unknown and compliance with diet is not satisfactory in PKU adults. A Previously established technique called indicator amino acid oxidation (IAAO) will be used to determine protein requirements from amino acid based formula vs. glycomacropeptide (GMP) in adults with PKU (≥ 19y). This study will help treat adults with enough protein ensuring maintenance of health.

ELIGIBILITY:
Inclusion Criteria:

-Adults more than 19 years of age who are diagnosed with PKU and clinically stable with no acute illness

Exclusion Criteria:

* Adults with PKU under age 19 year
* Adults diagnosed with PKU but are currently ill with a fever or cold

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
13 Co2 production | 8 hours (1 study day). 3 samples will collected as a baseline prior to isotope protocol and 6 samples after 2 hours and 30 minutes of starting the tracer protocol. Data will be reported an average of 2 years.
  Breath samples will be collected during the study to measure the rate of oxidation of tracer in the expired breath.
Lysine flux | 8 hours (1 study day). 1 sample will collected as a baseline prior to isotope protocol and 2 samples after 2 hours and 30 minutes of starting the tracer protocol. Data will be reported an average of 2 years.
  Urine samples will be collected during the study to measure the flux enrichment in urine.

SECONDARY OUTCOMES:
Phenylalanine concentrations | One sample (at 6th meal) after starting of the tracer protocol. Data will be reported an average of 2 years.
  Phenylalanine concentrations will be measured in blood.
Tyrosine concentrations | One sample (at 6th meal) after starting of the tracer protocol. Data will be reported an average of 2 years.
  Tyrosine concentrations will be measured in blood.
16 other amino acids | One sample (at 6th meal) after starting of the tracer protocol. Data will be reported an average of 2 years.
  16 other amino acids will be measured in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — BC Children's Hospital Research Institute, University of British Columbia; Sandra Sirrs, MD, Study Chair — University of British Columbia; Sylvia Stockler, MD, Study Chair — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada